CLINICAL TRIAL: NCT00114075
Title: Impact of Gait Analysis on Surgical Outcomes
Brief Title: Effects of Walking Analysis on Surgical Outcomes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5R01HS014169 (AHRQ); 5R01HS014169 (AHRQ)
Record Dates: First submitted 2005-06-13; First posted 2005-06-14 (Estimated); Last update posted 2012-07-18 (Estimated); Status verified 2011-08

CONDITIONS: Cerebral Palsy
Keywords: gait; walking; orthopedic surgery; orthopaedic surgery
MeSH Terms: conditions — Cerebral Palsy | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gait analysis (Experimental): Gait analysis report is available for treatment planning
  Interventions: Procedure: Surgery with gait analysis report
- Control (Active Comparator): Subject has gait analysis test, but report is not available for treatment planning
  Interventions: Procedure: Surgery without gait analysis report

INTERVENTIONS:
Procedure: Surgery with gait analysis report — Orthopaedic surgery with access to gait analysis report
  Arms: Gait analysis
Procedure: Surgery without gait analysis report — Orthopaedic surgery without access to gait analysis report
  Arms: Control

SUMMARY:
The purpose of this study is to evaluate the effects of pre-operative gait analysis testing on surgical outcomes in children with cerebral palsy who have problems walking.

DETAILED DESCRIPTION:
Gait analysis testing has been used to assist orthopaedic surgeons in developing treatment plans for children with gait abnormalities, particularly children with cerebral palsy. Previous studies have shown that gait analysis testing significantly impacts surgical decision-making for these patients. However, no controlled studies have been done to determine whether gait analysis and the subsequent changes in surgical decision-making affect clinical outcomes. Consequently, the use of gait analysis in clinical practice remains controversial. The purpose of this study is to conduct a randomized controlled trial to assess the effects of preoperative gait analysis on surgical outcomes in ambulatory children with cerebral palsy.

Comparison: Surgery with information from gait analysis testing compared with surgery without information from gait analysis testing.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cerebral palsy
* Able to walk
* Under evaluation for orthopedic surgery to correct walking problem(s)

Exclusion Criteria:

* Orthopaedic surgery in past 1 year
* Injection of botulinum toxin in past 6 months

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 186 (Actual)
Dates: Start 2005-01; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Change in walking ability at 1 year | 1 year
Change in walking efficiency at 1 year | 1 year

SECONDARY OUTCOMES:
Change in gross motor function at 1 year | 1 year
Change in quality of life at 1 year | 1 year
Additional treatment needed at 1 year | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Tishya AL Wren, Ph.D., Principal Investigator — Children's Hospital Los Angeles
Locations (2):
- United States (2):
  - Shriners Hospital for Children, Los Angeles, Los Angeles, California
  - Childrens Hospital Los Angeles, Los Angeles, California

REFERENCES:
- [Background] Kay RM, Dennis S, Rethlefsen S, Reynolds RA, Skaggs DL, Tolo VT. The effect of preoperative gait analysis on orthopaedic decision making. Clin Orthop Relat Res. 2000 Mar;(372):217-22. doi: 10.1097/00003086-200003000-00023. PMID 10738430
- See also: Agency for Healthcare Research and Quality — http://www.ahrq.gov/
- See also: United Cerebral Palsy — http://www.ucp.org/
- See also: Gait and Clinical Movement Analysis Society — http://www.gcmas.org/